CLINICAL TRIAL: NCT01087359
Title: Antiinflammatoric and Antioxidative Effect of Melatonin in Human Endotoxaemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Mahdi Alamili, MA
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: H-2-2010-010
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2010-10

CONDITIONS: Human Endotoxaemia
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- LPS + melatonin night (Active Comparator)
  Interventions: Drug: Melatonin
- LPS + placebo night (Placebo Comparator)
  Interventions: Drug: Melatonin
- LPS + melatonin day (Active Comparator)
  Interventions: Drug: Melatonin
- LPS + placebo day (Placebo Comparator)
  Interventions: Drug: Melatonin
- LPS night (Experimental)
  Interventions: Drug: Melatonin
- LPS day (Experimental)
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — 100 mg melatonin is tested on human endotoxaemia administrated on night and day time compared to placebo

SUMMARY:
This is a double blinded, randomised, crossover study with 12 healthy men between 18 and 40 year. The design is based on 6 days:

* day 1: On day time administration of LPS.
* day 2: On night time administration of LPS.
* day 3: On day time administration of LPS + Placebo.
* day 4: On day time administration of LPS + melatonin.
* day 5: On night time administration of LPS + placebo.
* day 6: On night time administration og LPS + melatonin.

Measuring the inflammatoric and oxidative response of LPS and the effect of melatonin compared to placebo on the endotoxaemia.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Age 18-49 year.
* Healthy
* No sleepiness disorders.
* No medication
* ASA I

Exclusion Criteria:

* Allergia to melatonin
* Women
* Smoking.
* Alcohol abuse.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Inflammatoric markers | measured before and after the administration of LPS endotoxin.
  IL-6 TNF-alpha YKL-40
Oxidative markers | measured before and after the administration of LPS endotoxin.
  Vit C MDA (malondialdehyde)

SECONDARY OUTCOMES:
Secondary outcome | constant measurment
  Holter Fatigue Karolinska Sleepness scale Blood pressure Heart rate Temperature

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Herlev, Denmark